CLINICAL TRIAL: NCT02892981
Title: Dead Space Evaluation During Exercise in Patients With Pulmonary Hypertension
Brief Title: Dead Space Evaluation in Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, Piergiuseppe Agostoni, Professor, Centro Cardiologico Monzino
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ccm257
Record Dates: First submitted 2016-06-10; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

ARMS (1):
- Pulmonary hypertension patients (Other): All Pulmonary hypertension patients enrolled in the study underwent a cardiopulmonary exercise test and hypoxia and hypercapnia tests
  Interventions: Other: cardiopulmonary exercise test,hypoxia and hypercapnia test

INTERVENTIONS:
Other: cardiopulmonary exercise test,hypoxia and hypercapnia test — class I and IV Pulmonary hypertension patients in stable haemodynamic status and optimized medical therapy underwent cardiopulmonary test and hypoxia and hypercapnia tests to evaluate the chemoreceptor sensitivity

SUMMARY:
Aim of the study is to evaluate the role of chemoreceptor activity and ventilation perfusion mismatch on the genesis of exercise induced hyperventilation in Pulmonary hypertension patients. So the investigators tested the chemoreceptor response at rest, both with hypoxic and hypercapnic stimuli, and the ventilatory response during exercise analyzing its two components, alveolar and dead space ventilation.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 and ≤ 80 years
* ability to understand the research protocol and willing to sign the study informed consent
* diagnosis of pulmonary arterial hypertension belonging to Class I and IV
* stable haemodynamic status and optimized medical treatment since at least 2 months
* ability to perform maximal cardiopulmonary exercise test and pulmonary diffusing capacity for carbon monoxide evaluation

Exclusion Criteria:

* relevant comorbidities
* usual contraindications for cardiopulmonary exercise test
* pulmonary hypertension associated to left heart and pulmonary disease, congenital heart diseases with evident cardiac shunts.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
dead space ventilation (measured in L/min) | 1 week
  Dead space ventilation is calculated through the equation: VT* [1- (863*VCO2)/(VE*PaCO2)], where VT = tidal volume, VCO2= CO2 output, VE= pulmonary ventilation,PaCO2 is the arterial partial pressure of CO2 and 863 is a constant.

SECONDARY OUTCOMES:
peripheral response to hypoxia (measured in L/min/O2) | 1 week
  the hypoxic test is based on the transient hypoxia (the patient inhales a mixture of nitrogen for 2-8 breaths, for 10-15 times); pulmonary ventilation (VE) and arterial oxygen saturation (O2 Saturation) by peripheral pulse oximetry is measured. The chemoreceptor sensitivity value is calculated as the slope of the trend line built on the two maximum consecutive VE and minimum O2 Saturation of each test.
peripheral response to hypercapnia (measured in L/min/mmHg) | 1 week
  the peripheral response to hypercapnia is evaluated through the single-breath technique (the patient inhales a mixture of 13% CO2 in air for a single breath); pulmonary ventilation (VE) and end-expiratory CO2 fraction (FetCO2) are measured and then they will be used to calculate the peripheral chemoreceptor sensitivity.In fact, the sensitivity of the chemoreceptor is calculated using the following formula VEs-VEc / (FetCO2s-FetCO2c) * (PB-47), where s and c indicate the data collected after hypercapnic stimulus and those collected during control air breathing ,respectively; PB is the atmospheric pressure in mmHg
central hypercapnic chemosensitivity (measured in L/min/mmHg) | 1 week
  the evaluation of the central response to hypercapnia is made through the re-breathing technique (the patient breathes through a reservoir containing 7% CO2 and 93% O2 for 4 minutes); pulmonary ventilation (VE) and partial pressure of end-tidal carbon dioxide (PetCO2) are evaluated. The slope of the curve describing the relationship between VE and PetCO2 identifies the central chemoreceptor sensitivity

REFERENCES:
- [Derived] Farina S, Bruno N, Agalbato C, Contini M, Cassandro R, Elia D, Harari S, Agostoni P. Physiological insights of exercise hyperventilation in arterial and chronic thromboembolic pulmonary hypertension. Int J Cardiol. 2018 May 15;259:178-182. doi: 10.1016/j.ijcard.2017.11.023. PMID 29579597